CLINICAL TRIAL: NCT02927028
Title: The Effects of Mastication and Digestion on the Bio Accessibility of Energy From Walnuts
Brief Title: The Effects of Mastication on Energy Release From Walnuts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 055-042
Record Dates: First submitted 2015-10-14; First posted 2016-10-06 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: energy availability; walnuts
MeSH Terms: conditions — Obesity | interventions — Mastication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chewing group (Other): 50 individuals, both male and female, between the ages of 18 and 60 years old, with a BMI between 18-35 kg/m2 from any ethnic/racial background will be recruited. Participants must have natural dentition and rate the hedonic value of all study foods between 3 and 7 on a 9-point category scale.
  Interventions: Other: Chewing

INTERVENTIONS:
Other: Chewing — On the first visit, the random nut treatments will include chewing walnuts, almonds and pistachios. The chewing conditions will include: 1) 5 g nuts alone, 2) 5 g nuts with 5 ml water, 3) 5 g nuts with 5 ml apple juice, 4) 5 g nuts with 5 g plain yogurt, 5) 5 g nuts with 5 g sweet yogurt.
  On visits 2 and 3 the treatments of either 28 g of walnuts or walnut butter will be presented.

SUMMARY:
With an emphasis on oral processing, this study seeks to characterize the mechanisms that account for the high satiation properties of walnuts and low energy yield during digestion.

DETAILED DESCRIPTION:
Recent evidence indicates up to 20% of the energy from walnuts is not absorbed. This low bio accessibility is comparable to almonds with markedly different physical properties and much higher than for pistachios with similar physical characteristics. These counter-intuitive findings require mechanistic explanations so they may be accepted and used to formulate policy and clinical recommendations. It is proposed that the differences in the structure of nuts accounts for the energy yield results. In addition, the whole nut yields superior effects on fullness and this leads to focus on oral processing. It may be that the mechanical act of chewing generates satiety sensations or it may be that the mechanical disruption of the parenchymal call walls releases lipid and protein and their higher concentrations activate the release of gut peptides associated with satiety.

Visit 1: Participants will report the Laboratory of Sensory and Ingestive Studies following and overnight fast, and having refrained from using oral care products for at least two hours prior to the visit. Participants who meet the BMI requirements, will have electrodes placed on their wrist, upper, and lower jaw and will be asked to chew the following stimuli: walnuts, almonds and pistachios for 15 seconds and expectorate the bolus into a beaker. However, when presented with 5 g walnuts participants will be asked to chew until the point where they would normally swallow and then spit the bolus into a beaker. The chewing conditions are randomized and include: 1) 5 g nuts alone, 2) 5 g nuts with 5 ml water, 3) 5 g nuts with 5 ml apple juice, 4) 5 g nuts with 5 g plain yogurt, 5) 5 g nuts with 5 g sweet yogurt. Following each chewing condition, participants will rate hedonic preference on a 9-point scale.

Visit 2 and 3: Following an overnight fast, the participant will be placed in a semi-supine position and a catheter will be placed in a vein in the antecubital space of one arm. A 9 ml baseline blood sample will be collected. Participants will complete a validated appetite questionnaire on a palm pilot right after the baseline blood draw. The participants will then consume 28 g of walnuts or 28 g walnut butter given in random order. Additional blood samples and appetite questionnaire will be taken at 15, 30, 45, 60,120, and 180 minutes. The blood will be stored in a minus 80 freezer to be analyzed at a later date for insulin, glucose, GLP-1, Ghrelin, and PYY.

ELIGIBILITY:
Inclusion Criteria:

* Natural dentition and no oral pathology
* Rate hedonic value of all study foods between 3 and 7 on a 9-point category scale.

Exclusion Criteria:

* BMI between 18-35 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Effects of oral processing on the energy yield from walnuts. | 7 months
  Released fat concentration following chewing.

SECONDARY OUTCOMES:
Particle size disruption | 7 months
  The proportion of particle size distributions of chewed samples (nuts) will be determined by sieving the boluses.

OTHER OUTCOMES:
Cell staining and counting | 7 months
  Quantify the effects of mastication on nut cell structure by quantify cell viability measured by cell size and number.
Appetite ratings | 7 months
  The effects of walnut consumption on fullness sensations will be measured using 100 mm visual analogue scale. Participants will rate their fullness after consuming 28 g of walnuts in two forms.
In vitro digestion | 7 months
  Released fat concentration following gastric and intestinal digestion.
Insulin | 7 months
  Blood samples will be taken an analyzed for insulin.
Glucose | 7 months
  Blood samples will be taken an analyzed for glucose.
GLP-1 | 7 months
  Blood samples will be taken an analyzed for GLP-1.
Ghrelin | 7 months
  Blood samples will be taken an analyzed for Ghrelin.
PYY | 7 months
  Blood samples will be taken an analyzed for PYY.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided